CLINICAL TRIAL: NCT02280434
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CBP-307 Following Oral Single and Multiple Escalating Dose Administration
Brief Title: Phase 1 Study Accessing the Safety and Tolerability of CBP-307
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry); Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-307AU001
Record Dates: First submitted 2014-10-20; First posted 2014-10-31 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBP-307 (Active Comparator): Participants will receive a single dose or once daily dose of CBP-307 for 28 days.
  Interventions: Drug: CBP-307
- Placebo (Placebo Comparator): Participants will receive a single dose or once daily dose of matching placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBP-307
  Arms: CBP-307
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of CBP-307 following oral single and multiple escalating dose administration in healthy subjects.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of CBP-307 following oral single and multiple escalating dose administration in healthy subjects. The study will have two parts: Part 1 will assess 5 dose levels of the drug in single dosing; and Part 2 will evaluate 3 dose levels in 28-day repeat dosing. The effect of food will also be evaluated in a single dosing study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained in writing for all subjects at enrollment into the study
* Healthy male subjects age between 18 and 55 years, inclusive
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive
* No clinically significant findings in the medical history and physical examination, especially with regard to the liver and gastrointestinal systems
* No clinically significant laboratory values and urinalysis, unless the investigator considers any abnormality to be clinically irrelevant
* Normal ECG, blood pressure, and heart rate, unless the investigator considers any abnormality to be clinically irrelevant
* Resting heart rate ≥ 55 bpm

Exclusion Criteria:

* Family history of premature CHD (Coronary Heart Disease)
* Any condition requiring the regular use of any medication
* Exposure to prescription medications or to drugs known to interfere with metabolism of drugs within 30 days prior to screening
* Exposure to any other medication, including over-the counter medications, herbal remedies and vitamins 14 days prior to randomization (except paracetamol (see Section 5.2 Prior and concomitant treatments)
* Participation in another study with any investigational drug in the 2 months preceding the study
* Treatment in the previous 3 months with any drug known to have a well defined potential for toxicity to a major organ
* Positive urine cotinine result at screening
* Be in the exclusion period of any previous study with investigational drugs
* Symptoms of a clinically significant illness in the 3 months before the study
* Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease
* Hemorrhoids or anal diseases with regular or recent presence of blood in feces
* History of significant allergic disease (e.g. medications) and acute phase of allergic rhinitis in the previous 2 weeks before randomization or any food allergy
* Blood or plasma donation of more than 500 ml during the previous 2 month before randomization and/or more than 50 ml in the 2 weeks prior to screening
* Subjects at risk for tuberculosis (TB), specifically subjects with: Current clinical, radiographic or laboratory evidence of active TB; history of active TB unless there is documentation that the prior anti-TB treatment was appropriate in duration and type;latent TB which has not been successfully treated; a positive quantiFERON® test at screening or within 6 months prior to Day 1
* Known positive test for HIV
* Known positive test for hepatitis B (antigens HBs, antibody HBc) or C, unless caused by immunization
* History of shingles or recurrent episodes of HSV1 or HSV2 infections
* Current evidence of drug abuse or history of drug abuse within one year before randomization
* History of alcohol abuse or active alcoholism as defined in Appendix A Definition of alcohol abuse
* Mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study
* Adults under guardianship and people with restriction of freedom by administrative or legal decisions
* Unlikely to comply with the clinical study protocol; e.g. uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Systolic blood pressure less than 95 mmHg or greater than 140 mmHg, or diastolic blood pressure less than or equal to 50 mmHg or greater than or equal to 95 mmHg.
* Subjects with resting heart rate less than 55 beats per minute or greater than 90 beats per minute.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 6 weeks
  Safety measurements will include vital signs, hematology, blood chemistry, blood pressure and other readouts.

SECONDARY OUTCOMES:
Plasma Concentrations of Study Drug Over Time and Maximal Plasma Concentration (Cmax) | Up to 6 weeks
Elimination Half-live (T1/2) of Study Drug | Up to 6 weeks
Exposure to Study Drug Measured as Area Under the Curve (AUC) | Up to 6 weeks
Effect of Study Drug on Blood Lymphocyte Counts | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, PhD, FRACP, Principal Investigator — Nucleus Network; Zheng Wei, PhD, Study Director — Suzhou Connect Biopharmaceuticals
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Lickliter J, Yang X, Guo J, Pan W, Wei Z. Icanbelimod (CBP-307), a next-generation Sphingosine-1-phosphate receptor modulator, in healthy men: pharmacokinetics, pharmacodynamics, safety, and tolerability in a randomized trial in Australia. Front Immunol. 2024 Jun 17;15:1380975. doi: 10.3389/fimmu.2024.1380975. eCollection 2024. PMID 38953034